CLINICAL TRIAL: NCT01176513
Title: GE148-002: A Phase 2, Open-label, Single-Center, Study to Assess GE-148 (18F) Injection Positron Emission Tomography(PET) Imaging to Detect Localized Prostate Cancer
Brief Title: GE-148-002: A Phase 2, Open-label, Single-Center Study to Assess GE-148 (18F) Injection PET Imaging to Detect Localized Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Subject enrollment
Sponsor: GE Healthcare (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-148-002; 10-C-0179; NCT01313091 (obsolete NCT alias)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; MRI; PET; GE-148 (18F)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GE 148-002 (Experimental)
  Interventions: Drug: GE-148 (18F)

INTERVENTIONS:
Drug: GE-148 (18F) — All subjects will receive an i.v. dose of GE-148 (18F) Injection at 10 mCi (370 MBq) to provide adequate image quality throughout the specified imaging period.
  Other Names: GE-148 (18F) Injection

SUMMARY:
Background:

- GE-148 (18F) is a new drug that is designed to attach to prostate cancer cells. Researchers are interested in combining the drug with a small amount of radioactive material to allow prostate cancer lesions to appear more clearly on imaging scans. Researchers are also interested in determining whether the combination can help make cancer cells in pelvic lymph nodes easier to detect through imaging studies. GE-148 (18F) will be used to examine individuals who are scheduled to have surgery on their prostate cancer.

Objectives:

- To evaluate the effectiveness of GE-148 (18F) in detecting prostate cancer and cancer cells in pelvic lymph nodes using positron emission tomography and magnetic resonance imaging scanning.

Eligibility:

- Men at least 18 years of age who have been diagnosed with prostate cancer and are scheduled to have prostate removal surgery.

Design:

* Participants will be screened with a physical examination, medical history, blood tests, and imaging studies.
* Participants will have magnetic resonance imaging (MRI) and positron emission tomography (PET) scans with GE-148 (18F) prior to their scheduled surgery. The MRI and PET scans may be performed on the same day or on different days, depending on the schedule set by the study researchers.
* Tissue samples taken during prostate removal surgery, including prostate tissue and pelvic lymph nodes, will be collected for further study of the effectiveness of GE-148 (18F).

DETAILED DESCRIPTION:
Background:

* Accurate imaging of prostate cancer is important for developing targeted minimally invasive therapies
* GE-148 (18F) Injection is a drug product formulation known as [18F]FACBC which is a synthetic leucine amino acid analogue. Preliminary studies demonstrated efficacy in primary prostate cancer and metastatic/recurrent prostate cancers. We propose to evaluate GE-148 (18F) Injection as a PET radiopharmaceutical for the detection of prostate cancer.

Objectives: Primary Objective:

* To differentiate the magnitude of uptake and retention of GE-148 (18F) Injection between malignant prostate tumors, non-malignant prostate pathology, and regions of normal prostate tissue in subjects with prostate cancer.
* To assess the safety of a single dose of GE-148 (18F) Injection in subjects with prostate cancer.

Secondary Objectives:

* To assess the relationship between the magnitude of uptake of GE-148 (18F) Injection with quantitative assessment of AAT expression in malignant prostate tumors, non-malignant prostate pathology, and regions of normal prostate tissue.
* To assess the relationship between the magnitude of uptake of GE-148 (18F) Injection with quantitative assessment of Ki-67 expression in malignant prostate tumors, non-malignant prostate pathology, and regions of normal prostate tissue.
* To assess the relationship between the magnitude of uptake of GE-148 (18F) Injection in malignant prostate tumors and their Gleason Score.
* To assess the ability of GE-148 (18F) Injection to detect the number of discrete malignant prostate tumors confirmed by histopathology.
* To assess the relationship between the magnitude of uptake of GE-148 (18F) Injection with quantitative measurement of AAT and Ki-67 expression in pelvic lymph nodes showing uptake of GE-148 (18F) Injection, where available.
* To compare the ability of PET/CT imaging with GE-148 (18F) Injection to predict prostate malignancy and distinguish it from other pathologies (inflammation, hyperplasia, atrophy, hemorrhage) with that of T2W MRI, DCE MRI, MR DWI, and MRSI performed at 3T.

Eligibility:

* Subject is 18 years old, ECOG 0-2, with documented prostate cancer (minimum 1 core).
* Subject must be scheduled to undergo standard of care prostatectomy at NIH CC

Serum creatinine within 2 weeks prior to MRI less than or equal to1.8mg/dl, estimated GFR(eGFR) must be greater than 30 ml/min/1.73m2.

-Chemistry parameters: Aspartate aminotransferase (AST), Alanine transferase (ALT)2 x of the upper limits of normal; total bilirubin, of less than 2 x the upper limits of normal or less than 3.0 mg/dl in patients with Gilbert's syndrome.

Design:

Thirty subjects with localized prostate cancer scheduled for prostatectomy will undergo dynamic GE-148 (18F) Injection PET/CT imaging, and undergo a standard-of-care endorectal coil/pelvic multiparametric MRI . Results will be compared with pathology.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subject is male and is greater than or equal to 18 years old.
* Subject must be scheduled to undergo standard of care prostatectomy for presumed localized prostate cancer at the NIH Clinical Center.
* Recent (within 12 months of study entry but not within 8-12 weeks before start of imaging study) prostate biopsy indicating the presence of adenocarcinoma of the prostate gland in which at least sextant biopsies were obtained.
* Subjects must have a minimum of 1 positive-for-cancer biopsy core.
* Serum creatinine within 2 weeks prior to MR imaging less than or equal to 1.8 mg/dl and eGFR must be greater than 30 ml/min/1.73m(2)
* Chemistry parameters: AST and ALT 2 x of the upper limits of normal; total bilirubin, of less than or equal to 2 x the upper limits of normal or less than 3.0 mg/dl in patients with Gilbert's syndrome.
* Eastern Cooperative Oncology Group (ECOG) Performance score of 0 to 2.
* Ability to provide informed consent. All subjects must sign an informed consent form indicating their understanding of the investigational nature and risks of the study before any protocol-related studies are performed.
* The subject has a clinically acceptable medical history, physical examination and vital signs findings during the screening period (from within 21 days before administration of GE-148 (18F) Injection).

EXCLUSION CRITERIA:

* Known allergy to gadolinium.
* Subjects for whom participating would significantly delay the scheduled standard of care therapy.
* Subjects with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results.
* Subjects with severe claustrophobia unresponsive to oral anxiolytics.
* Subjects with contraindications to MRI

  * Subjects weighing more than 136 kg (weight limit for scanner table).
  * Subjects with pacemakers, cerebral aneurysm clips, shrapnel injury, or other implanted electronic devices or metal not compatible with MRI.
* Subjects with contraindication to endorectal coil placement

  * Severe hemorrhoids.
  * Surgically absent rectum.
* Other medical conditions deemed by the principle investigator (or associates) or sponsor to make the subject ineligible for protocol procedures.
* Subjects who have previously received radiation therapy to the pelvis.
* Subjects who have received androgen-deprivation therapy.
* The subject has received, or is scheduled to receive, another IMP from 1 month before to 1 week after administration of GE-148 (18F) Injection.
* Subjects with chronic renal failure (eGFR less than 30 ml/min/1.73m(2)).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gordon, PhD, Study Director — GE Healthcare
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jung JA, Coakley FV, Vigneron DB, Swanson MG, Qayyum A, Weinberg V, Jones KD, Carroll PR, Kurhanewicz J. Prostate depiction at endorectal MR spectroscopic imaging: investigation of a standardized evaluation system. Radiology. 2004 Dec;233(3):701-8. doi: 10.1148/radiol.2333030672. PMID 15564406
- [Background] Swindle P, Eastham JA, Ohori M, Kattan MW, Wheeler T, Maru N, Slawin K, Scardino PT. Do margins matter? The prognostic significance of positive surgical margins in radical prostatectomy specimens. J Urol. 2005 Sep;174(3):903-7. doi: 10.1097/01.ju.0000169475.00949.78. PMID 16093984
- [Background] el-Gabry EA, Halpern EJ, Strup SE, Gomella LG. Imaging prostate cancer: current and future applications. Oncology (Williston Park). 2001 Mar;15(3):325-36; discussion 339-42. PMID 11301831
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2010-C-0179.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 25 subjects were enrolled in this study and 3 subjects withdrew prior to dosing with this product. As a result, 22 subjects were used in the analysis for this study.
Groups:
- GE 148-002: GE-148 (18F) : All subjects will receive an i.v. dose of GE-148 (18F) Injection at 10 mCi (370 MBq) to provide adequate image quality throughout the specified imaging period.
Period: Overall Study
Arm/Group | GE 148-002
Started | 25
Completed | 22
Not Completed | 3
Not completed — Withdrew subjects prior to dosing | 3

BASELINE CHARACTERISTICS:
Population: 25 subjects were enrolled in the study and 3 subjects withdrew prior to dosing with the product. As a result, 22 subjects were used in the analysis.
Arm/Group | GE 148-002
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (6.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Magnitude of Uptake and Retention of GE-148 (18F) Injection in Malignant Prostate Tumors, Non-malignant Prostate Pathology, and Regions of Normal Prostate Tissue in Subjects With Prostate Cancer, Using PET/CT Imaging.
Description: Quantitative measurements of the level of uptake of GE-148 (18F) Injection into each tissue type (malignant prostate tumors, non-malignant prostate pathology, and regions of normal prostate) calculated as Standardized Uptake Values (SUVs), using histopathology as the standard of truth.
Time Frame: After GE-148 (18F) Injection administration.
Population: Efficacy analyses were not performed because GE Healthcare terminated the study early for administrative reasons.
Groups:
- GE 148-002: GE-148 (18F) : All subjects will receive an i.v. dose of GE-148 (18F) Injection at 10 mCi (370 MBq) to provide adequate image quality throughout the specified imaging period.
  Efficacy analyses were not performed because GE Healthcare terminated the study early for administrative reasons.
Arm/Group | GE 148-002
Number analyzed (Participants) | 0

2. Secondary Outcome: To Compare the Ability of PET/CT Imaging With GE-148 (18F) Injection to Predict Prostate Malignancy and Distinguish it From Other Pathologies (Inflammation, Hyperplasia, Atrophy, Hemorrhage) With That of T2W MRI, DCE MRI, MR DWI, and MRSI Performed at 3T.
Description: Use of descriptive statistics to compare the ability of the PET/CT imaging and MRI to predict malignancy, based on histopathology as the standard of truth, on a subject basis and per lesion basis.
Time Frame: After GE-148 (18F) Injection administration
Population: Efficacy analyses were not performed because GE Healthcare terminated the study early for administrative reasons.
Arm/Group | GE 148-002
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | GE 148-002
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 2/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GE 148-002 (N=22)
Dysgeusia (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No